CLINICAL TRIAL: NCT05531682
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 2 Study to Evaluate the Efficacy and Safety of Different Dosing Regimens of HB0017 Injection in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: A Study to Evaluate the Efficacy and Safety of HB0017 in Patients With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huabo Biopharm Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0017-05
Record Dates: First submitted 2022-08-31; First posted 2022-09-08 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2022-09

CONDITIONS: Plaque Psoriasis
Keywords: HB0017; Chronic Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Experimental: HB0017 dosing regimen 1 (Experimental): HB0017 low dose short intervals of subcutaneous injection
  Interventions: Drug: HB0017
- Experimental: HB0017 dosing regimen 2 (Experimental): HB0017 low dose long intervals of subcutaneous injection
  Interventions: Drug: HB0017
- Experimental: HB0017 dosing regimen 3 (Experimental): HB0017 high dose long intervals of subcutaneous injection
  Interventions: Drug: HB0017
- Placebo Comparator: placebo group (Placebo Comparator): Placebo was subcutaneously injected into the 12 weeks turnover HB0017 subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Subjects will receive several injections of Placebo
  Arms: Placebo Comparator: placebo group
Drug: HB0017 — Subjects will receive HB0017 in different dosing regimens
  Other Names: HB0017 dosing regimens
  Arms: Experimental: HB0017 dosing regimen 1; Experimental: HB0017 dosing regimen 2; Experimental: HB0017 dosing regimen 3

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multi-center Phase 2 study to evaluate the efficacy and safety of HB0017 in subjects with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multi-center Phase 2 study to evaluate the efficacy and safety of HB0017 in subjects with moderate to severe plaque psoriasis. The study will consist of 3 periods: up to 5 weeks screening period, 28 weeks treatment period, 8 weeks Safety Follow-Up period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent
* Diagnosis of chronic plaque psoriasis with or without psoriatic arthritis for at least 6 months prior to Screening
* Psoriasis Area and Severity Index(PASI)>=12 and body surface area(BSA) >=10% and static Physician's Global Assessment (sPGA) score 3 or greater on a 5-point scale
* Candidates for systemic psoriasis therapy and/or phototherapy and/or chemo phototherapy
* Women who are at childbearing age(not pregnant or breast-feeding), and subjects and their partners voluntarily use contraceptive methods deemed effective by the investigator during treatment and for at least 6 months after the last study medication

Key Exclusion Criteria:

* Forms of psoriasis other than chronic plaque psoriasis.
* History or evidence of active tuberculosis, Patients with evidence of latent tuberculosis may enter the trial after sufficient treatment according to protocol.
* Positive results of confirmatory serology test for hepatitis B, hepatitis C, HIV or syphilis at screening.
* History of a serious or systemic infection within 4 weeks before screening.
* History of malignancy of any organ system within the past 5 years.
* Inadequate washout period for prior drug therapy.
* Previous use of secukinumab, ixekizumab or any other drug that targets Interleukin 17( IL-17) or IL-17 receptor.
* Any medical conditions, in the opinion of the Investigator or the Sponsor's medical monitor, would place the subject at risk, interfere with study participation or study results interpretation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
PASI 90 response | Week 12
  Proportion of subjects who achieve Psoriasis Area and Severity Index (PASI) 90 response or higher at week 12
sPGA 0/1 response | Week 12
  Proportion of subjects who achieve static Physician Global Assessment (sPGA) 0 or 1

SECONDARY OUTCOMES:
PASI 75 response | Week 12
  Proportion of subjects who achieve PASI 75 response or higher
Adverse events | From baseline through 36 weeks
  Treatment Related Adverse events (TEAEs)/serious adverse events (SAEs)
Immunity | From baseline through 36 weeks
  Number and proportion of subjects who developed anti-drug antibodies (ADAs) Following Study Treatment
PK characteristics | From Baseline through 36 weeks
  Population pharmacokinetics (PK), Apparent Total Clearance (CL/F)， Apparent Volume of Distribution (V/F) of HB0017
PASI responses up to 36 Weeks | From Baseline through 36 weeks
  Proportion of subjects who achieve PASI 50, PASI 75, PASI 90 , PASI 100 response up to 36 weeks
sPGA 0/1 up to 36 Weeks | From Baseline through 36 weeks
  Proportion of subjects who achieve
PD characterestics | From Baseline through 36 weeks
  HB0017 concentrations in serum at different time points
PASI score change | From Baseline through 36 weeks
  change in PASI From Baseline to Week 36
Percent change in PASI | From Baseline through 36 weeks
  Percent change in PASI From Baseline to Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong zhang, Principal Investigator — Peking University People's Hospital
Locations (21):
- China (21):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of Wannan Medical College, Wuhu, Anhui
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The first hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Dermatology Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Shandong Provincial Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Skin Disease Hospital of Shandong First Medical University, Jinan, Shandong
  - Yantai Yuhuangding hospital, Yantai, Shandong
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Third People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Shanghai Skin Disease Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No